CLINICAL TRIAL: NCT03766828
Title: Dialysis Catheter Placement in Patients With Thoracic Central Venous Occlusion
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Guerkan SENGOELGE, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Other Study IDs: Vienna-DialysisAccess
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Central Venous Catheter Thrombosis
Keywords: thoracic central venous occlusion; Dialysis access
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inside-out-access technique with inside-out access device
  Interventions: Procedure: inside-out-access technique with inside-out access device (Surfacer (R))
- access technique including Sharp recanalization
  Interventions: Procedure: access technique including Sharp recanalization

INTERVENTIONS:
Procedure: inside-out-access technique with inside-out access device (Surfacer (R)) — inside-out-access technique with (Surfacer (R)) with a new CE certified device (Surfacer (R), Bluegrass Vascular)
  Groups: inside-out-access technique with inside-out access device
Procedure: access technique including Sharp recanalization — access technique with Sharp recanalization via interventional radiology
  Groups: access technique including Sharp recanalization

SUMMARY:
A unique inside-out-access technique with a new CE certified device (Surfacer (R) Bluegrass Vascular, San Antonio, Tx, USA) enables repetitive and confident right-sided placement of central venous catheters in hemodialysis patients with thoracic central venous occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic central venous occlusion

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with thoracic central venous occlusion requiring vascular access
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Achievement of dialysis access | 1 day

SECONDARY OUTCOMES:
procedure related complications | 3 months
  infections, bleeding, hematoma or pericardial effusions and intervention related parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Sengölge, Principal Investigator — Department of Medicine III, Division of Nephrology
Locations (1):
- Department of Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Vienna, Austria